CLINICAL TRIAL: NCT06287437
Title: A Single-center, Double-blinded, Randomized, Placebo-controlled Trial to Evaluate the Effectiveness and Safety of Low-frequency Injection of HRS9531 in Control of Weight Regain in Obese Subjects With and Without Diabetes
Brief Title: HRS9531 Controls Weight Regain in Obese Subjects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Study Principal Investigator, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2023-335R
Record Dates: First submitted 2024-01-02; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The subjects receive sequential once weekly and low frequency subcutaneous injection of HRS 9531
  Interventions: Drug: HRS9531
- Control (Placebo Comparator): The subjects receive low frequency subcutaneous injection of the placebo
  Interventions: Drug: HRS9531 placebo

INTERVENTIONS:
Drug: HRS9531 — HRS9531 escalated to the protocol-specified dose once weekly injection for 24 weeks ，then low frequency injection for 12 weeks.
  Arms: Intervention
Drug: HRS9531 placebo — HRS9531 placebo low frequency injection for 12 weeks.
  Arms: Control

SUMMARY:
This is a single-center, double-blinded, randomized, placebo-controlled phase II study to explore the effectiveness, safety and energy balance mechanism of low-frequency continuous subcutaneous injection of HRS9531 to inhibit weight regain in obese non-diabetic and obese diabetic patients

ELIGIBILITY:
Inclusion Criteria:

1. 30-60 years old, female and male.
2. BMI:30-40kg/m2.
3. Non diabetes or type 2 diabetes with HbA1c between 7-10%.

Exclusion Criteria:

1. Weight change ≤5 kg within 3 months.
2. Hb<110g/L.
3. Serum triglycerides 5.7 mmol/L.
4. Impaired liver function ：ALT or AST≥3×ULN，TB≥2×ULN.
5. Impaired renal function：eGFT < 45 ml/min.
6. Hemodiastase or Serum lipase≥3×ULN.
7. TSH>6.0 mIU/L or<0.4 mIU/L.
8. Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg.
9. lth Questionnaire-9 (PHQ-9) score ≥15.
10. Type 1 diabetes.
11. Proliferative diabetic retinopathy, ketoacidosis or hyperglycemia hypertonic state within 3 months.
12. In the investigator's judgment, there were circumstances that affected subject safety or otherwise interfered with the evaluation of results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Body Weight from 24 weeks | 36 weeks
  Percentage change in body weight from the low-frequency injection phase for HRS9531 compared with placebo

SECONDARY OUTCOMES:
Energy intake change from 24 weeks | 24-36 weeks
  Differences in energy intake changes between the HRS9531 group and the placebo group from week36-week24
Energy expenditure change from 24 weeks | 24-36 weeks
  Differences in energy expenditure changes between the HRS9531 group and the placebo group from week36-week24
Metabolic adaptation from 24 weeks | 24-36 weeks
  Differences in metabolic adaptation changes between the HRS9531 group and the placebo group from week36-week24（Metabolic adaptation=Actual measured resting energy expenditure-Predicted resting energy expenditure. The Actual measured resting energy expenditure will be measured using the Maastricht Instruments Room Calorimeter ADVANCE. The predicted energy expenditure will be fitted by multiple linear regression according to the age, sex, and body composition information of the subjects at baseline.）
Systolic blood pressure and diastolic blood pressure change from 24 weeks | 24-36 weeks
  Differences in systolic blood pressure and diastolic blood pressure changes between the HRS9531 group and the placebo group from week36-week24
Body fat rate change from 24 weeks | 24-36 weeks
  Differences in body fat rate changes between the HRS9531 group and the placebo group from week36-week24
Serum total cholesterol change from 24 weeks | 24-36 weeks
  Differences in Serum total cholesterol changes between the HRS9531 group and the placebo group from week36-week24
Triglyceride change from 24 weeks | 24-36 weeks
  Differences in Triglyceride changes between the HRS9531 group and the placebo group from week36-week24
Nonestesterified fatty acid change from 24 weeks | 24-36 weeks
  Differences in nonestesterified fatty acid changes between the HRS9531 group and the placebo group from week36-week24
Energy intake at baseline | 0 weeks
  Differences in energy intake at baseline in obese diabetic subjects, relative to obese non-diabetic subjects.
Energy expenditure at baseline | 0 weeks
  Differences in energy expenditure at baseline in obese diabetic subjects, relative to obese non-diabetic subjects.
Appetite at baseline (assessed by Visual Analogue Scale subjective rating scale) | 0 weeks
  Differences in appetite at baseline in obese diabetic subjects, relative to obese non-diabetic subjects (Appetite was assessed using the Visual Analogue Scale subjective rating scale. On a standard scale of 100mm in length, the left end (0mm) means "not at all" and the right end (100mm) means "extremely").
Percent Change in Body Weight at 24 weeks | 24 weeks
  Obese diabetic subjects, relative to obese non-diabetic subjects, difference in body weight change after once weekly injection of HRS9531
Appetite at 24 weeks (assessed by Visual Analogue Scale subjective rating scale) | 24 weeks
  Obese diabetic subjects, relative to obese non-diabetic subjects, difference in appetite after once weekly injection of HRS9531(Appetite was assessed using the Visual Analogue Scale subjective rating scale. On a standard scale of 100mm in length, the left end (0mm) means "not at all" and the right end (100mm) means "extremely").
Energy expenditure at 24 weeks | 24 weeks
  Obese diabetic subjects, relative to obese non-diabetic subjects, difference in energy expenditure after once weekly injection of HRS9531
Energy intake at 24 weeks | 24 weeks
  Obese diabetic subjects, relative to obese non-diabetic subjects, difference in Energy intake after once weekly injection of HRS9531

OTHER OUTCOMES:
Change of body weight at 24 weeksl from baseline | 24 weeks
  Change of body weight from baseline to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Zhongshan Hosptial, Fudan University
Locations (1):
- Xiaoying Li, Shanghai, China